CLINICAL TRIAL: NCT05432453
Title: Investigation of the Relationship Between Functional Constipation and Sacroiliac Joint Dysfunction
Brief Title: The Relationship Between Functional Constipation and Sacroiliac Joint Dysfunction
Status: Recruiting | Type: Observational
Sponsor: Abant Izzet Baysal University (Other)
Responsible Party: Principal Investigator, Ömer Osman Pala, Assistant Professor, Abant Izzet Baysal University
Other Study IDs: AIBU-FTR-BI-2
Record Dates: First submitted 2022-06-21; First posted 2022-06-27 (Actual); Last update posted 2024-02-12 (Actual); Status verified 2024-02

CONDITIONS: Constipation - Functional; Sacroiliac Joint Somatic Dysfunction
Keywords: constipation; women; rehabilitation
MeSH Terms: conditions — Constipation

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Weeks
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Women with constipation: Bowel functional markers (defecation frequency, defecation time, and stool density) and constipation-related quality of life of women with constipation will be evaluated with the Constipation Severity Scale, Constipation Quality of Life Scale, 7-day bowel diary, and Bristol Stool Scale.
  Sacroiliac joint dysfunctions of women with constipation will be evaluated by standing forward bending test, sitting forward bending test, compression test, posterior friction test and Patrick-Faber test.
- Women without constipation (Control): Bowel functional markers (defecation frequency, defecation time, and stool density) and constipation-related quality of life of women without constipation will be evaluated with the Constipation Severity Scale, Constipation Quality of Life Scale, 7-day bowel diary, and Bristol Stool Scale.
  Sacroiliac joint dysfunctions of women without constipation will be evaluated by standing forward bending test, sitting forward bending test, compression test, posterior friction test and Patrick-Faber test.

SUMMARY:
The purpose of this study; to compare individuals with and without chronic constipation in terms of sacroiliac joint dysfunction and to examine the relationship between chronic constipation and sacroiliac joint.

DETAILED DESCRIPTION:
Constipation is a heterogeneous, polysymptomatic and multifactorial disease. Many symptoms are used to define the term constipation, such as hard stool, excessive straining, few bowel movements, use of digital maneuvers during defecation, abdominal bloating, and a feeling of inadequate evacuation.

Chronic constipation is seen in approximately 14% of the world. It is seen on average 2 times more in women.

Visceral and somatic neural control of defecation is provided by the Sacral 2-4 segments of the spinal cord. It is in neural relationship with the sacroiliac joint and pelvic floor muscles, which also provide innervation from the same segments. These visceral and somatic structures can affect each other through viscerosomatic and somatovisceral reflexes. This means that an afferent input from the rectum can reflect on and around the sacroiliac joint.

Based on this connection, we think that primary chronic constipation without an organic cause may be associated with sacroiliac joint dysfunction. In the literature review, no study examining this relationship was found.

This study is planned to evaluate individuals with and without chronic constipation in terms of sacroiliac joint dysfunction and to examine the relationship between chronic constipation and sacroiliac joint.

ELIGIBILITY:
Inclusion Criteria (for functional constipation group):

* Voluntary participation in the research
* Fulfill the diagnostic criteria for functional constipation (Rome IV)
* Being women
* Not using laxatives for at least the last 4 weeks

Inclusion Criteria (for control group):

* Voluntary participation in the research
* Being women
* Not having functional constipation

Exclusion Criteria:

* Having cooperation problems
* Being pregnant
* Being breast-feeding
* Taking medication for depression, hypertension, sleep disorders, and pain
* Having parkinson, stroke, spinal cord injury, multiple sclerosis, hypothyroidism, Diabetes Mellitus, cerebral Palsy, thyroid problems, cancer, presence of tumor, presence of hernia, endometriosis, neuropathy, myopathy, scleroderma, inflammatory bowel diseases (Crohn, gastrointestinal tuberculosis, celiac, colon diverticulum, colonoscopy), cognitive impairment
* Having neurological or metabolic or malignant disorders
* Having a history of open abdominal surgery
* Having a history of pelvic and abdominal radiotherapy

Ages: 18 Years to 65 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes
Study Population: Functional constipation criteria (Rome IV) will be use for functional constipation group.
  1. Must include 2 or more of the following:
  1. Straining during more than one-fourth (25%) of defecations
  2. Lumpy or hard stools (BSFS 1-2) more than one-fourth (25%) of defecations
  3. Sensation of incomplete evacuation more than one-fourth (25%) of defecations
  4. Sensation of anorectal obstruction/blockage more than one-fourth (25%) of defecations
  5. Manual maneuvers to facilitate more than one fourth (25%) of defecations (e.g., digital evacuation, support of the pelvic floor)
  6. Fewer than three spontaneous bowel movements per week 2. Loose stools are rarely present without the use of laxatives 3. Insufficient criteria for irritable bowel syndrome
Sampling Method: Non-Probability Sample
Enrollment: 128 (Estimated)
Dates: Start 2022-05-16 (Actual); Primary Completion 2024-05-01 (Estimated); Study Completion 2024-05-01 (Estimated)

PRIMARY OUTCOMES:
The Standing Forward Bend Test (One of Sacroiliac Joint Dysfunction Tests) | one day
  The participant stands with their feet shoulder-width apart. The physiotherapist places the thumbs on the participant's posterior superior iliac spine. The physiotherapist stands or kneels behind the participant with their eyes aligned with the posterior superior iliac spine. The participant is instructed to lean forward, trying to touch their fingers. The forward bending movement should be done without bending the knees and in a way that does not cause pain.
  The standing forward bending test gives information about whether there is a blockage in one of the sacroiliac joints and if there is a blockage, on which side it is. At the end of the movement, the test is positive on the anterior side of the spina iliaca posterior superior. In the positivity of this test, the forward bending test in sitting is performed to distinguish between iliac and sacrum dysfunction.
The Sitting Forward Bend Test (One of Sacroiliac Joint Dysfunction Tests) | one day
  The participant sits with their legs slightly apart. The physiotherapist stands or kneels behind the participant with their eyes aligned with the posterior superior iliac spine and palps the posterior superior of the spina iliaca. The participant is asked to lean forward as far as possible without pain. If at the end of the movement the asymmetry in the posterior superior spina iliaca becomes more pronounced than in the foot, it is defined as a dysfunction of the sacrum, less pronounced than that of the foot, or a dysfunction of the ilium if absent.
The Compression Test (One of Sacroiliac Joint Dysfunction Tests) | one day
  The participant lies on their side with their hips flexed to 45° and knees flexed to 90°. The physiotherapist stands behind the participant and applies pressure over the iliac crest to the contralateral iliac crest. The test is applied to the other side as well. Pain caused by compression makes the test positive.
The Posterior Friction Test (One of Sacroiliac Joint Dysfunction Tests) | one day
  Axial pressure is applied across the femur, bringing the hip of the participant in the supine position to 90° flexion and adduction of the femur. The occurrence of pain suggests a pathology in the sacroiliac joint.
The Patrick Faber Test (One of Sacroiliac Joint Dysfunction Tests) | one day
  The ipsilateral hip and knee joint of the participant in the supine position is flexed, and the heel is placed on the opposite knee. The physiotherapist provides stabilization over the contralateral spina iliaca anterior superior to maintain the neutral position. The test stresses the anterior sacroiliac ligaments and hip joint. The test is considered positive with pain occurring in the sacroiliac joint area.
7-day bowel diary | one week
  Individuals will be asked to complete a bowel diary for 7 days for evaluation. Individuals will be asked to mark each day they defecate, how long they stay in the toilet at each defecation, mark if there is a feeling of incomplete emptying, note the changes in nutrition and fluid consumption and drug use, and record their stool consistency by looking at the Bristol stool scale.

SECONDARY OUTCOMES:
The Constipation Severity Scale | one day
  Constipation severity of individuals will be evaluated with the Constipation Severity Scale.
  star_border The Constipation Severity Scale is a scale to determine the frequency, density and difficulty/difficulty of individuals during defecation. There are 16 questions in the scale.The lowest total score that can be obtained from the constipation severity scale is 0, and the highest is 73. A high score from the scale indicates that the symptoms are serious.
The Constipation Quality of Life Scale | one day
  This scale consists of 28 items and consists of "physical discomfort" (questions 1-4), "psychosocial discomfort" (questions 5-12), "worry/anxiety" (questions 13-23) and "satisfaction" (questions 24-28). It has 4 subdomains. The answer options for the scale questions are in the five-point Likert scale type and the item scores range from 1 to 5. The lowest score that can be obtained from the scale is 28, and the highest score is 140. Higher scores on the scale mean that quality of life is more negatively affected.

CONTACTS AND LOCATIONS:
Overall Officials: Ömer Osman Pala, Principal Investigator — Bolu Abant İzzet Baysal University
Locations (1):
- Faculty of Health Sciences Bolu Abant İzzet Baysal University, Bolu, Turkey (Türkiye)